CLINICAL TRIAL: NCT04415489
Title: SIS Versus Office Hysteroscopy for Uterine Cavity Evaluation Prior to IVF: a Randomized Control Trial
Brief Title: SIS Versus Office Hysteroscopy for Uterine Cavity Evaluation Prior to IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-3077
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Results first posted 2021-04-14 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-03

CONDITIONS: Infertility
Keywords: Assisted Reproduction
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial comparing satisfaction between saline infusion sonography and office hysteroscopy for screening evaluation of the uterine cavity prior to embryo transfer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Office Hysteroscopy (Active Comparator): Use of office hysteroscope with operative port to evaluate uterine cavity, and potentially treat minor abnormalities within the same procedure with hysteroscopic graspers. This involve inserting the hysteroscope through the cervix and instillation of saline for a direct look at the cavity.
  Interventions: Device: Office hysteroscopy
- Saline Infusion Sonography (SIS) (No Intervention): This is our institution's current first line approach for screening evaluation of the uterine cavity. If not enrolled in the study, patients are required to do this to move forward with embryo transfer. It involves instillation of saline into the uterus via a small catheter with simultaneous imaging with pelvic ultrasound.

INTERVENTIONS:
Device: Office hysteroscopy — Use of hysteroscopy in the clinical setting to directly visualize the cavity. If pathology amenable to immediate treatment is visualize, removal will be attempted by hysteroscopic graspers.
  Other Names: LiNA OperaScope
  Arms: Office Hysteroscopy

SUMMARY:
Saline infusion sonography (SIS) and hysteroscopy are commonly employed methods for uterine cavity evaluation. While hysteroscopy is regarded as the gold standard for diagnosis of intra-uterine pathology, it is not often used as an initial screening tool because of provider concerns about in-office tolerability, operating room costs, and use of anesthesia. The investigators aim to compare SIS and office hysteroscopy with respect to patient and provider satisfaction. Additionally, the investigators aim to assess the capability of office-based hysteroscopy to manage intra-uterine pathology at the time of diagnosis and reduce delays and supernumerary procedures.

DETAILED DESCRIPTION:
Saline infusion sonography (SIS) and hysteroscopy are commonly employed methods for uterine cavity evaluation. SIS is often performed as a screening tool in the office for uterine evaluation since it is straight-forward to perform, well-tolerated has low overhead cost. If uterine pathology is suspected on SIS, subsequent hysteroscopy is typically performed in the operating room. Hysteroscopy remains the gold standard for diagnosis of intra-uterine pathology and offers the opportunity for intervention at time of diagnosis, but often is not used as the initial screening tool because of provider concerns about in-office tolerability, equipment cost and maintenance. Technology advancements, however, has introduced an affordable, disposable, small caliber hysteroscopes with an operative channel to make it possible for this type of assessment to be performed in the office setting with the addition of a 'see and treat' modality. If used to perform initial uterine cavity evaluation, hysteroscopy may offer expedited diagnosis, treatment, and avoidance of general anesthesia. If superior specificity is demonstrated, it may also lower the false positive rate, preventing unnecessary delays to a patient's projected treatment plan, and unnecessary exposure to anesthesia risks. To date, no randomized control trials have compared the satisfaction of patients and providers to saline infusion sonography versus office hysteroscopy without anesthesia in initial cavity evaluation with the ability to immediately address intra-uterine pathology.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 - 50
* Patients undergoing routine cavity evaluation for planned in vitro-fertilization cycles

Exclusion Criteria:

* Clinical or radiologic suspicion of intrauterine pathology including myomas, severe intrauterine adhesions or retained products of conception
* Those with medical criteria not suitable office hysteroscopy due to requirement of advanced tools or preparation not available in the office such as history of bleeding disorder or medical co-morbidity

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Moustafa, MD, Principal Investigator — University of North Carolina, Chapel Hill; Linnea Goodman, MD, Study Chair — University of North Carolina, Chapel Hill
Locations (1):
- UNC Fertility, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 9 months and ending 3 years following article publication.
Access Criteria: Investigator proposing to use data has IRB, IEC, or REB approval and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Moustafa S, Rosen E, Goodman L. Patient and provider satisfaction with saline ultrasound versus office hysteroscopy for uterine cavity evaluation prior to in vitro fertilization: a randomized controlled trial. J Assist Reprod Genet. 2021 Mar;38(3):627-634. doi: 10.1007/s10815-021-02065-9. Epub 2021 Feb 1. PMID 33527249

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Office Hysteroscopy | Saline Infusion Sonography (SIS)
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Office Hysteroscopy | Saline Infusion Sonography (SIS) | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (4.6) | 34.7 (4.9) | 34.3 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 3 | 1 | 4
  Race/Ethnicity: Black or African American | 5 | 6 | 11
  Race/Ethnicity: White | 42 | 39 | 81
  Race/Ethnicity: Hispanic | 0 | 4 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] — Population: BMI data were missing for 5 participants in the SIS arm.
  Kg/m^2
    number analyzed (Participants) | 50 | 45 | 95
    (all) | 26.2 (6.4) | 27.7 (6.4) | 26.9 (6.4)
Infertility Diagnosis [Count of Participants; unit: Participants]
  Diminished ovarian reserve | 3 | 7 | 10
  Endometriosis | 3 | 1 | 4
  Ovulatory dysfunction | 10 | 7 | 17
  Male factor | 17 | 10 | 27
  Tubal factor | 1 | 4 | 5
  Unexplained | 10 | 13 | 23
  Other | 6 | 8 | 14
Prior Uterine Surgery [Count of Participants; unit: Participants]
  Dilation and curettage | 4 | 9 | 13
  Myomectomy | 4 | 2 | 6
  Polypectomy | 0 | 2 | 2
  Lysis of adhesions | 0 | 0 | 0
  Caesarean section | 7 | 7 | 14
  Other | 1 | 0 | 1
  None | 34 | 30 | 64
History of Uterine Pathology [Count of Participants; unit: Participants]
  History of uterine pathology | 2 | 4 | 6
  No history of uterine pathology | 48 | 46 | 94
Vaginal Delivery History [Count of Participants; unit: Participants]
  Prior Vaginal Delivery | 9 | 11 | 20
  No prior Vaginal Delivery | 41 | 39 | 80
Number of Participants with Prior Cervical Surgery [Count of Participants; unit: Participants] | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction
Description: Survey with Likert scale administered to record patients overall satisfaction during their procedure. Scoring range is 1-5, with 1 corresponding Very Unsatisfied (worse) and 5 corresponding to Very Satisfied (better).
Time Frame: Immediately following imaging modality (less than 30 minutes)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Office Hysteroscopy | Saline Infusion Sonography (SIS)
Number analyzed (Participants) | 50 | 50
units on a scale | 4.92 (0.34) | 4.84 (4.7)
Statistical Analysis 1: Comparison: Office Hysteroscopy vs Saline Infusion Sonography (SIS); Test type: Superiority; p = 0.57, Fisher Exact — The a priori threshold for statistical significance was p < 0.05

2. Primary Outcome: Pain Scores
Description: Survey administered to record patients pain scores during their procedure. Score range is 1-10, with one being minimal pain (better) and 10 being the worst pain ever experienced (worse).
Time Frame: Immediately following imaging modality (less than 30 minutes)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Office Hysteroscopy | Saline Infusion Sonography (SIS)
Number analyzed (Participants) | 50 | 50
units on a scale | 3.38 (1.85) | 2.44 (1.64)
Statistical Analysis 1: Comparison: Office Hysteroscopy vs Saline Infusion Sonography (SIS); Test type: Superiority; p < 0.01, t-test, 2 sided — The a priori threshold for statistical significance was p < 0.05

3. Primary Outcome: Provider Satisfaction
Description: Survey with Likert scale administered to record providers overall satisfaction during their procedure. Scoring range is 1-5, with 1 corresponding Very Unsatisfied (worse) and 5 corresponding to Very Satisfied (better).
Time Frame: Immediately following imaging modality (less than 30 minutes)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Surveys analyzed
Arm/Group | Office Hysteroscopy | Saline Infusion Sonography (SIS)
Number analyzed (Participants) | 2 | 5
Number analyzed (Surveys analyzed) | 50 | 50
units on a scale | 4.76 (0.69) | 4.56 (0.81)
Statistical Analysis 1: Comparison: Office Hysteroscopy vs Saline Infusion Sonography (SIS); Test type: Superiority; p = 0.11, Fisher Exact — The a priori threshold for statistical significance was < 0.05

4. Secondary Outcome: Time to Complete
Description: Length of time to complete procedure in minutes
Time Frame: During the allotted procedure only
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Office Hysteroscopy | Saline Infusion Sonography (SIS)
Number analyzed (Participants) | 50 | 50
minutes | 4.61 (2.42) | 3.98 (2.03)
Statistical Analysis 1: Comparison: Office Hysteroscopy vs Saline Infusion Sonography (SIS); Test type: Superiority; p = 0.16, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05

5. Secondary Outcome: Number of Patients Requiring Secondary Procedure
Description: Number of patients requiring a secondary procedure, either for management of pathology or inability to complete initial procedure.
Time Frame: Through study completion, up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Office Hysteroscopy | Saline Infusion Sonography (SIS)
Number analyzed (Participants) | 50 | 50
Participants | 1 | 11
Statistical Analysis 1: Comparison: Office Hysteroscopy vs Saline Infusion Sonography (SIS); Test type: Superiority; p < 0.01, Fisher Exact — The a priori threshold for statistical significance was < 0.05

6. Secondary Outcome: Time to Infertility Treatment
Description: Number of days to achieve planned fertility treatment
Time Frame: Through study completion, up to 1 year
Population: Number of Patients requiring secondary procedure was used instead to represent potential for treatment delay. This measure was abandoned and no data was collected, based on the following factors making it less reliable: (1) variability of ability to add a second procedure case on the same day (for patient and/or provider), and (2) presence of other uncontrollable factors contributing to fertility treatment delay
Arm/Group | Office Hysteroscopy | Saline Infusion Sonography (SIS)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Positive Predictive Value of SIS
Description: Number of Participants with SIS Findings, Validated by Subsequent Hysteroscopy
Time Frame: Through study completion, up to 1 year
Population: Reported for those participants with abnormal finding during SIS procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Saline Infusion Sonography (SIS)
Number analyzed (Participants) | 11
Participants | 9

8. Secondary Outcome: Ability to Manage Pathology With Office Hysteroscopy
Description: Number of participants with pathology on hysteroscopy successfully managed within same procedure
Time Frame: During the allotted procedure only
Population: Participants with abnormal finding during office hysteroscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Office Hysteroscopy
Number analyzed (Participants) | 17
Participants | 16

9. Post Hoc Outcome: Number of Participants With Pathology Found
Description: Descriptive characterization of pathology identified for participants, if any, during procedure.
Time Frame: During the allotted procedure only
Measure: Count of Participants; unit: Participants
Arm/Group | Office Hysteroscopy | Saline Infusion Sonography (SIS)
Number analyzed (Participants) | 50 | 50
Participants
  Polyps | 10 | 7
  Myoma | 0 | 1
  Adhesions | 2 | 2
  Retained product | 5 | 1
  Uterine anomaly | 2 | 0
  Inconclusive | 0 | 1
  None | 31 | 38
Statistical Analysis 1: Comparison: Office Hysteroscopy vs Saline Infusion Sonography (SIS); Test type: Superiority; p = 0.12, Fisher Exact — The a priori threshold for statistical significance was < 0.05

ADVERSE EVENTS:
Time Frame: From the time of office procedure through 30 days afterwards.
Arm/Group | Office Hysteroscopy | Saline Infusion Sonography (SIS)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT04415489/Prot_SAP_000.pdf